CLINICAL TRIAL: NCT07172074
Title: Improving Vaccine Outcomes in Older Adults-Quantitative
Brief Title: Comparing Relative Strengths of Statistical Associations Between Psychological Traits and Vaccination-Related Outcomes I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Aaron Scherer, Associate Professor of Internal Medicine, University of Iowa
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 202211127; 5K01AG065440 (NIH)
Record Dates: First submitted 2025-09-03; First posted 2025-09-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Vaccination; Vaccination Hesitancy; Vaccination Promotion; Psychological Aspects
Keywords: Vaccination; Vaccine Confidence; Attitudinal Roots; Psychological Traits; Motivated Social Cognition
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Decades of research has shown that information is sought out, evaluated, and used in a biased way in order to satisfy people's motivations to satisfy their psychological needs. This bias in information processing is broadly referred to as "motivated social cognition". Three general psychological needs people are motivated to satisfy include:
  1. Managing threats: Motivations to eliminate perceived physical, emotional, or ideological threats
  2. Reducing uncertainty: Motivations to reduce uncertainty, complexity, ambiguity, or disorder
  3. Achieving social goals: Motivations for relationships with like-minded others and keeping groups distinct I propose that different forms of these motives may underlie vaccine outcomes and the processing of vaccine-related information.
Who Masked: Participant, Investigator
Masking Description: Randomization was done by the online survey platform (Qualtrics)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Planned Missingness Design Block A (Experimental): Respondents were randomized to complete one of three blocks (items predetermined by being randomized to blocks, with 1/3 of items in each block) of the psychological trait measures
  Interventions: Diagnostic Test: General Psych Trait Measure; Other: Vaccine-Specific Psych Trait Measures
- Planned Missingness Design Block B (Experimental): Respondents were randomized to complete one of three blocks (items predetermined by being randomized to blocks, with 1/3 of items in each block) of the psychological trait measures
  Interventions: Diagnostic Test: General Psych Trait Measure; Other: Vaccine-Specific Psych Trait Measures
- Planned Missingness Design Block C (Experimental): Respondents were randomized to complete one of three blocks (items predetermined by being randomized to blocks, with 1/3 of items in each block) of the psychological trait measures
  Interventions: Diagnostic Test: General Psych Trait Measure; Other: Vaccine-Specific Psych Trait Measures

INTERVENTIONS:
Diagnostic Test: General Psych Trait Measure — Respondents were randomized to answer whether psychological trait questions were general or about vaccines
Other: Vaccine-Specific Psych Trait Measures — Respondents were randomized to answer whether psychological trait questions were general or about vaccines

SUMMARY:
The goal of this study was to identify psychological motives that had the strongest statistical associations with vaccine outcomes in order to identify novel intervention targets to be used in vaccine promotion efforts. A national sample of US adults completed an online survey containing a variety of vaccine-related measures and psychological trait measures.

DETAILED DESCRIPTION:
A national sample of US adults were recruited through Dynata, an online survey panel company, to complete an online survey. Participants completed a variety of vaccine-related survey items and an unprecedented number (>20) of psychological trait measures. This was possible by using a Planned Missingness Design, where respondents only answer a predetermined subset of survey questions, which allows us to include more measures without significantly increasing the burden for participants.

Participants were randomized to one of the three question blocks, where each block had a predetermined set of items that were roughly 1/3 of the items from each psychological trait measure. They were also randomized to complete questions that were about the psychological traits in general or about vaccines specifically.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate
* Agree to provide quality responses

Exclusion Criteria:

* Quota completed (Equal #s of respondents in each group)

  * Age group: 18-49, 50-64, 65+
  * Race/ethnicity: Non-Hispanic White, Non-Hispanic Black, Hispanic
  * Income: <$50K, $50K or more
  * Gender: Female, Male or other gender identity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1786 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Vaccine attitudes | Day 1
  Feelings towards vaccines on a 7-point scale, with Very negative (1) and Very positive (7) as the scale anchors
Vaccination History | Day 1
  Indicated if they had received up to 7 age-recommended vaccines (Response options: No, Yes, Don't know/Unsure)

SECONDARY OUTCOMES:
Psychological trait measures | Day 1
  26 measures: Needle phobia, Disgust sensitivity, Distrust, Conspiratorial mindset, Medical ambiguity aversion, Open-minded thinking, Self-protection motivation, Psychological reactance, 7 Moral Foundations, Self-construal, Social dominance orientation, Misinformation susceptibility, Faith in intuition, Delay discounting, Outcome bias, Scientific knowledge, Subjective numeracy, Health literacy, Medical maximizing-minimizing, Emotional reactivity to rare events
7C Antecedents to Vaccination | Day 1
  Single item to measure each antecedent to vaccination
Attitudes towards Complementary and Alternative Medicine | Day 1
  6 item measure
Personal Characteristics/Demographics | Day 1
  16 characteristics: Gender, Age, Race/ethnicity, Income, State of residence, Zip code, Relationship status, Education, Work in medical field, Economic political ideology, Social political ideology, Political party affiliation strength, Religiosity, Religious ideology, Subjective health, Health conditions

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Scherer, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be available upon request or posted on Dr. Scherer's personal Open Science Foundation website (https://osf.io/wgf4j)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately
Access Criteria: Anyone will be able to access any of the study materials and/or date upon request or if posted to Dr. Scherer's OSF website (https://osf.io/wgf4j)